CLINICAL TRIAL: NCT00327717
Title: A Multicenter, Placebo-controlled, Double-blind Study to Evaluate the Efficacy and Safety of Zonisamide in the Treatment of Partial Seizures
Brief Title: Evaluating the Efficacy and Safety of Zonisamide in the Treatment of Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2090-AS086-311
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Partial Seizures
Keywords: Epilepsy; Partial seizures
MeSH Terms: conditions — Seizures; Epilepsy | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Zonisamide 100 mg tablet (Experimental)
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — Patients entered a 4-week titration period, during which zonisamide dosing began at 100 mg/day for the first 2 weeks, increased to 200 mg/day for the 3rd week, and to 300 mg/day for the 4th week, reaching 300 mg/d at the end of the titration period. 300 mg/d was the target dose in the titration period and must be reached. Dose increment was continued to 400 mg/d if this was tolerated by the patient.
  Other Names: Zonegran
  Arms: Zonisamide 100 mg tablet
Drug: Placebo — Patients in placebo group were titrated with placebo in the same way as in zonisamide group.
  Arms: Placebo

SUMMARY:
The objectives of this trial are to evaluate the safety and efficacy of Zonisamide as adjunctive therapy in medically refractory patients receiving other antiepileptic drugs (AEDs).

ELIGIBILITY:
According to the International League Against Epilepsy (ILAE) classification of seizure type (1981) and international classification of epilepsies and epileptic syndromes (ILAE, 1989), definite diagnosis of partial seizures (with or without secondary generalized seizures) refractory to current anti epilepsy drug (AED) therapy.

Inclusion criteria:

1. Adult male or female, 16 to 70 years old;
2. Classified according to the ILAE classification of seizure type (1981) and international classification of epilepsy and epileptic syndromes (ILAE, 1989) into partial seizures (with or without secondary generalized seizures);
3. Based on the retrospective subject diary, at least 4 partial seizures per month ( 4 weeks ) within 12 weeks prior to entry;
4. No more than 8 secondary generalized tonic, clonic, or tonic-clonic seizures per month within 12 weeks prior to entry;
5. Antiepileptic therapy including at least 1-2 concomitant AEDs and were on a stable dose(s) of the same AEDs for the 3 months prior to enrollment;
6. Had performed electro encephalogram (EEG) within 6 months prior to entry, and computer tomography (CT) or magnetic resonance imaging (MRI) examination to mainly exclude space-occupying disease;
7. Was able to count seizure frequencies;
8. Women with child bearing potential, were not to be pregnant or nursing, and must have agreed to practice during the study a reliable form of contraception (oral contraceptive, condom, intrauterine device or diaphragm).
9. Signed written informed consent and agreed to comply with the protocol.

Exclusion criteria:

1. History or evidence of a progressive central nervous system (CNS) disease;
2. Nonepileptic seizures and pseudoepileptic seizures;
3. Severe mental retardation or unstable psychical status;
4. Clinically significant cardiac, hepatic, renal, or hematological disease, uncontrolled hypertension (systolic blood pressure (SBP) ≥150 and/or diastolic blood pressure (DBP) ≥100mmHg), Symptomatic ischemic heart disease, cerebral infarction or atherosclerosis obliterans;
5. History of malignant neoplastic disease;
6. Any condition that might interfere the pharmacokinetics (absorption, distribution, and/or excretion) of drugs, such as liver or kidney dysfunction, hypoproteinemia;
7. Glucose-6-phosphate dehydrogenase (G-6-PD) deficiency or history of hemolytic anemia or acute intermittent porphyria.
8. History of kidney stone;
9. History of alcohol or drug abuse within 2 years;
10. Sensitivity to sulfonamide medications or history of severe drug allergy;
11. Administration of monoamine oxidase inhibitor (MAOI), antidepressants or antipsychotic a psycho-tropic within 14 days prior to entry;
12. History of status epileptics in the past years or seizure clusters where individual seizures cannot be counted ;
13. History of zonisamide administration;
14. History of acetazolamide administration to treat epilepsy within 2 months prior to entry;
15. Joined the clinical trial of other AEDs within 30 days prior to entry;
16. Pregnant women or women in lactation;
17. Abnormal clinical laboratory values with clinical significance judged by investigators (for example, if abnormal hepatic function is caused by concurrent other AEDs, the abnormal value within 2 times of normal could be acceptable);
18. Inability of subject to return for scheduled visits or to comply with any other aspect of the protocol.
19. Subjects who, in the opinion of the investigator, were poor medical candidates or pose any other risk for therapy with an investigational drug.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Di Hong, Study Director — Eisai China Inc.
Locations (8):
- China (8):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking Union Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Hua-shan Hospital, Shanghai, Shanghai Municipality
  - XiÆan Xijing Hospital, XiÆan, Shanxi
  - Chengdu Huaxi Hospital, Chengdu, Sichuan

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide 100 mg Tablet: Patients entered a 4-week titration period, during which zonisamide dosing began at 100 mg/day for the first 2 weeks, increased to 200 mg/day for the 3rd week, and to 300 mg/day for the 4th week, reaching 300 mg/d at the end of the titration period. 300 mg/d was the target dose in the titration period and must be reached. Dose increment was continued to 400 mg/d if this was tolerated by the patient.
Period: Overall Study
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Started | 120 | 120
Completed | 111 | 106
Not Completed | 9 | 14
Not completed — Adverse Event | 6 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide 100 mg Tablet | Placebo | Total
Number analyzed (Participants) | 111 | 106 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.72 (12.18) | 30.69 (11.59) | 31.73 (11.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 43 | 97
  Male | 57 | 63 | 120
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 120 | 97 | 217
Region of Enrollment [Number; unit: participants]
  China | 111 | 106 | 217

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Change From Baseline in All Partial Seizure Frequency (Complex Partial Seizures (CP)+ Simple Partial Seizures (SP) + Secondary Generalization Seizures (SGS)) During the Fixed-dose Phase
Description: The median percent change in seizure frequency of all partial seizures (CP+SP+SGS) from baseline during the fixed-dose phase.
Time Frame: Baseline and 16 weeks
Population: Full analysis set (FAS)
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Percent Change | -48.42 (73.83) [-100 to 475] | -26.58 (157.22) [-100 to 1360.74]
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.028, ANOVA

2. Secondary Outcome: The Mean Percent Change From Baseline in Complex Partial (CP) Seizure Frequency
Description: The Mean Percent Change in seizure frequency of CP from baseline during the fixed-dose phase.
Time Frame: Baseline and 16 weeks
Population: FAS population. Complex partial seizure patients
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 69 | 69
Percent Change | -31.65 (87.28) | -25.21 (68.23)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.253, ANOVA

3. Secondary Outcome: The Mean Percent Change From Baseline in Simple Partial (SP) Seizure Frequency
Description: The Mean percent change in seizure frequency of SP from baseline during the fixed-dose phase.
Time Frame: Baseline and 16 weeks
Population: FAS Population. Simple partial seizure patients
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 29 | 25
Percent Change | -49.14 (62.06) | 56.03 (318.43)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.211, ANOVA

4. Secondary Outcome: The Mean Percent Change From Baseline in Partial Seizures With Secondary Generalization (SGS)
Description: The mean percent change in seizure frequency of SGS from baseline during the fixed-dose phase.
Time Frame: Baseline and 16 weeks
Population: FAS Population. Secondary generalization patients
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 36 | 42
Percent Change | -53.2 (54.81) | -4.08 (178.66)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.516, ANOVA

5. Secondary Outcome: Responder Rate
Description: Responder rate is defined as percentage of participants with >=50% reduction in seizure frequency from baseline.
Time Frame: Baseline and 16 weeks
Population: FAS Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Percentage of Participants | 48.6 | 34.9
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.044, X^2 test

6. Secondary Outcome: Mean Number of Seizure Free Days
Description: Mean number of seizure free days per 28 day period during fixed dose phase
Time Frame: 12 weeks
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Days | 22.31 (6.14) | 21.43 (7.07)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.090, X^2 test

7. Secondary Outcome: Mean Percentage of Change in Seizure Free Days
Time Frame: 16 weeks
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Percent Change | 79.69 (21.93) | 76.52 (25.26)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.090, X^2 test

8. Secondary Outcome: Mean Time to First Seizure (Days)
Description: Mean time to first seizure during fixed dose phase
Time Frame: 16 weeks
Population: FAS Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Days | 22.31 (6.14) | 21.43 (7.07)
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.162, X^2 test

9. Secondary Outcome: Percentage of Seizure-free Participants During Fixed-dose Phase
Description: Percentage of seizure-free participants during fixed-dose phase
Time Frame: 16 weeks
Population: FAS Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Percentage of Participants | 1.8 | 2.8
Statistical Analysis 1: Comparison: Zonisamide 100 mg Tablet vs Placebo; Test type: Superiority or Other; p = 0.678, X^2 test

10. Secondary Outcome: Drop - Out Rate
Description: Number of Participants who dropped out of the study. In the Study drop-out rate is defined as number of participants.
Time Frame: 16 weeks
Population: FAS Population
Measure: Number; unit: Number of Participants
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Number analyzed (Participants) | 111 | 106
Number of Participants | 4 | 6

ADVERSE EVENTS:
Description: Placebo group has 2 fewer subjects - consent withdrawn 1 and lost to follow up 1.
Arm/Group | Zonisamide 100 mg Tablet | Placebo
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/118
Other Adverse Events (participants affected / at risk) | 95/120 | 75/118
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide 100 mg Tablet (N=120) | Placebo (N=118)
Headache (Nervous system disorders) | 13 (16) | 6 (8)
Dizziness (Nervous system disorders) | 12 (15) | 13 (16)
Memory impairment (Nervous system disorders) | 8 (8) | 1 (1)
White blood cell count decreased (Investigations) | 10 (10) | 4 (4)
Platelet count decreased (Investigations) | 7 (7) | 4 (4)
Weight decreased (Investigations) | 6 (6) | 4 (4)
somnolence (Psychiatric disorders) | 15 (18) | 17 (18)
nausea (Gastrointestinal disorders) | 13 (14) | 7 (7)
Abdominal distention (Gastrointestinal disorders) | 6 (6) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 22 (22) | 6 (7)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 17 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No